CLINICAL TRIAL: NCT02684994
Title: Client-directed Cognitive Processing Therapy
Acronym: CPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Indianapolis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0619
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Trauma; Sexual assault; Sexual abuse; Physical assault; Physical abuse; PTSD; Interpersonal Violence; Women
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive Processing Therapy (Other): Cognitive Processing Therapy
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Cognitive-processing therapy is a well-supported treatment for reactions following traumatic events. It includes 12 individual psychotherapy sessions and consists of 4 components: education about trauma responses, experiencing emotions related to the assault, development of skills for examining the truth of thoughts, and examination of beliefs in areas commonly influenced by the trauma.
  Other Names: CPT; Client-directed CPT

SUMMARY:
This study will take place over approximately 6 months and includes 3 assessment appointments (where information will be gathered, but no direct treatment provided) and 12 treatment sessions of cognitive processing therapy if eligible.

DETAILED DESCRIPTION:
The purpose of this research study is to examine the effectiveness of a client-directed version of a well-supported psychological therapy, cognitive processing therapy (CPT), for the treatment of psychological effects of traumatic experiences. Participants in this study are expected to be women who have experienced one or more interpersonal violence experiences (i.e. physical or sexual assault).

During the first assessment, participants will be interviewed by a qualified investigator/interviewer. The investigator/interviewer will ask participants about life experiences and reactions, including traumatic experiences and symptoms participants might be experiencing. This portion of the study will take approximately 2-3 hours. If participant's assessment reveals that participant is eligible for the study participant will begin the treatment portion of the study. If eligible, participant will also be given a packet of questionnaires to complete before participant's first treatment session. If participant is not eligible for the study, investigator/interviewer will provide participant with a list of referrals from which participant could seek treatment with other agencies.

If participant begins the treatment portion of the study, participant will participate in a client-directed version of cognitive processing therapy (CPT). CPT is a treatment designed to help participant understand the ways participant's traumatic experience has affected various aspects of participant's life (feelings, beliefs, behaviors, etc.). The treatment will consist of four main components: education about trauma responses, experiencing emotions related to the assault, development of skills for examining the truth of thoughts, and examination of beliefs in areas commonly influenced by traumatic experiences. During this treatment, participant will be exploring the ways in which the assault has affected participant's beliefs, such as participant's beliefs about participant's own safety, trust, and ability to have relationships. In the sessions, participant will explore these areas to discover and change the ways participant believes, since the assault has led to feelings of distress, fear, anxiety, and depression. Participant will be asked to do activities in between sessions each week, which will ask participant to think and write about participant's traumatic experiences. The treatment includes 12 sessions, each for one hour. Sessions will be held once or twice a week. The current version of CPT will include all the components of the regular CPT treatment, but may vary in order of sessions. The regular treatment protocol provides sessions in a set order, but the current study will allow participant some choices in when participant complete certain activities.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years of age or over, experienced one or more interpersonal violence events, traumatic event happened over a month ago, no traumatic events in the last 3 months, must be proficient in English

Exclusion Criteria:

* Current psychosis, mania, active suicidal ideation; Substance use disorder in the last 6 months; in a relationship with perpetrator of violence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
change in PTSD symptoms | pre-treatment, post-treatment, 3 month follow-up
  Clinician administered clinical interview (Clinician Administered PTSD Scale) assessing PTSD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S Elwood, Ph.D., Principal Investigator — University of Indianapolis
Locations (1):
- University of Indianapolis, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT02684994/Prot_SAP_000.pdf